CLINICAL TRIAL: NCT04522206
Title: An Analysis of the Efficacy of a Pre-Emptive Multimodal Pain Regimen in Reducing Acute Post-Operative Pain and Narcotic Pain Medication Requirements in Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-00734
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Results first posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative; Spine Injuries and Disorders; Narcotic Use
MeSH Terms: conditions — Pain, Postoperative; Disease | interventions — Methylmalonic Acid; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: A prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients undergoing elective spine surgery (Experimental)
  Interventions: Drug: Pre-op Multimodal analgesia (MMA) regimen + standard post-op oxycodone

INTERVENTIONS:
Drug: Pre-op Multimodal analgesia (MMA) regimen + standard post-op oxycodone — The study subjects will be assigned to the defined pre-op MMA regimen with standard postop oxycodone based pain control regimen given on an as needed basis. The treatment group outcomes will be compared to patients outside of the study including a historical control group (receiving only post-op pain regimen) prior to the implementation of the new regimen. The studied treatment group will receive within 3 hours before surgery an oral MMA regimen consisting of:
  Acetaminophen 975 mg Celecoxib 200 mg Gabapentin 300 mg Oxycodone 10 mg Extended Release

SUMMARY:
The aim of this study is to investigate the hypothesis that multimodal pain regimen (consisting of acetaminophen, celecoxib, gabapentin, and oxycodone) administered pre-operatively before elective spine surgery significantly decreases acute pain post-operatively as well as decreasing requirements of post-op opioids for pain control in PACU as compared to patients undergoing elective spine surgery without a pre-operative pain regimen.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective spine surgery at NYU Winthrop
* Age over 18 years

Exclusion Criteria:

* History of neuromuscular disorders
* History of inflammatory arthropathies
* History of spine metastases or active cancer in spine
* Medical History including any of the following: renal dysfunction, gastric ulcers, hepatic dysfunction, coagulopathic/bleeding disorders, prior adverse or allergic reactions to any of the medications in the study
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tariq, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to the PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Undergoing Elective Spine Surgery
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing Elective Spine Surgery
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 36
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) for Pain
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Undergoing Elective Spine Surgery
Number analyzed (Participants) | 44
score on a scale | 4.8 (2.6)

2. Primary Outcome: Opioid Sparing and Rescue Time
Description: Time interval from patient extubation to time when pain medication is first demanded in the PACU
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Patients Undergoing Elective Spine Surgery
Number analyzed (Participants) | 44
Hours | 1.5 (2.2)

3. Secondary Outcome: Length of Stay in Hospital
Time Frame: Up to 12 days
Measure: Mean (Full Range); unit: Hours
Arm/Group | Patients Undergoing Elective Spine Surgery
Number analyzed (Participants) | 44
Hours | 139 [7 to 270]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patient self-reporting and office follow-ups
Arm/Group | Patients Undergoing Elective Spine Surgery
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT04522206/Prot_SAP_000.pdf